CLINICAL TRIAL: NCT00349986
Title: The Determination of the First Dose and the Optimal Time of Administration of Insulin Glargine Combined With Oral Antidiabetic Drug in Poorly Controlled Type II Diabetic Patients
Brief Title: LANTUSTITR: Insulin Glargine in Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: prematurely terminated due to loss of interest
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4059
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Insuline glargine

SUMMARY:
The rationale of the study is to determine:

* the first dose and the titration of basal insulin
* the exact daily time administration of basal insulin in poorly controlled type II diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Insufficient combined oral antidiabetic treatment (biguanide + sulfonylurea)
* BMI >25 kg/m2 , <30 kg/m2
* HbA1c value >7.0%, <9.0% within one month

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Known malignancy
* Drug or alcohol abuse
* Severe liver disease
* Renal failure (se Creatinine > 150 micro mol/l)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
HgbA1c measurement

CONTACTS AND LOCATIONS:
Overall Officials: László Erős, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Budapest, Hungary